CLINICAL TRIAL: NCT07196319
Title: "From One Problem to Another, Comparing the Incidence of Compensatory Hyperhidrosis After T3 Vs. T3-4 Sympathectomy"
Brief Title: "Incidence of Compensatory Hyperhidrosis After T3 Vs T3-4 Sympathectomy"
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelmoneim Ahmed, principal investigator, Assiut University
Other Study IDs: CH post T3 &T3-4 Sympathectomy
Record Dates: First submitted 2025-09-13; First posted 2025-09-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Compensatory Hyperhidrosis; Compensatory Sweating
Keywords: compensatory; hyperhidrosis; sympathectomy
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T3 sympathectomy: patients who underwent T3 sympathectomy for primary hyperhidrosis
- T3-4 sympathectomy: patients who underwent through T3-4 sympathectomy for primary hyperhidrosis

SUMMARY:
The goal of this study is to compare the proportion of compensatory hyperhidrosis patients after sympathectomy at T3 level and sympathectomy at T3-4 level. The main question it aims to answer is:

can sympathectomyv at one level decrease the incidence of compensatory hyperhidrosis after primary hyperhidrosis.

DETAILED DESCRIPTION:
Primary hyperhidrosis is a chronic condition characterized by excessive sweating beyond physiological needs, commonly affecting the palms, axillae, face, or soles. This disorder is largely attributed to neurogenic hyperexcitability within the sympathetic nervous system's pathways innervating the eccrine sweat glands.When conservative treatments such as topical agents or oral medications fail, endoscopic thoracic sympathectomy (ETS) is considered an effective surgical option. However, a major postoperative complication is compensatory hyperhidrosis (CH)-the development of excessive sweating in previously unaffected areas such as the trunk, back, or thighs. CH can significantly impact patient satisfaction and quality of life, often becoming more distressing than the original condition.

The extent and level of sympathectomy have been proposed as key factors influencing the incidence and severity of CH. While higher levels or multilevel resections (e.g., T2-4) are associated with increased rates of CH, more limited approaches such as T3-only resection are thought to reduce this risk. However, definitive evidence comparing T3 versus T3-4 sympathectomy remains limited and inconsistent across studies.

This study aims to compare the incidence and severity of compensatory hyperhidrosis following T3 versus T3-4 sympathectomy for primary hyperhidrosis. Understanding these differences may help refine surgical approaches to minimize CH and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary hyperhidrosis
* Patients with palmar and\or axillary hyperhidrosis.
* Age ≥ 6 years

Exclusion Criteria:

* History of Prior thoracic surgery.
* History of prior disorder that cause hyperhidrosis ( obesity,autonomic neuropathy,menopause,gout,etc…)
* History of prior systemic diseases cause hyperhidrosis (hyperthyroidism,DM,pheochromocytoma,Parkinson's disease,etc…)
* Patients with psychological problems.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: population of study are patients with primary hyperhidrosis who are going through T3 or T3-4 sympathectomy.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-25 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of compensatory hyperhidrosis following T3 versus T3-4 sympathectomy. | 1 year post-sympathectomy

SECONDARY OUTCOMES:
severity of Compensatory hyperhidrosis by hyperhidrosis disease severity scale | 1 year post sympathectomy
  1. The sweating is never noticeable and doesn't interfere with daily activities.
  2. The sweating is tolerable but sometimes interferes with daily activities.
  3. The sweating is barely tolerable and frequently interferes with daily activities.
  4. The sweating is intolerable and always interferes with daily activities.
recurrence rates of primary hyperhidrosis | 1 year post sympathectomy
site of compensatory hyperhidrosis | 1year post sympathectomy

REFERENCES:
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Strutton DR, Kowalski JW, Glaser DA, Stang PE. US prevalence of hyperhidrosis and impact on individuals with axillary hyperhidrosis: results from a national survey. J Am Acad Dermatol. 2004 Aug;51(2):241-8. doi: 10.1016/j.jaad.2003.12.040. PMID 15280843
- [Background] 4. Lin TS, et al. Clinical experience of thoracoscopic sympathetic block for primary hyperhidrosis: analysis of 3450 cases. J Thorac Cardiovasc Surg. 2001;121(3):566-74.
- [Background] 3. Hussein AF, et al. Unilevel (T3) versus Bilevel (T3 - T4) Sympathictomy in the Management of Palmar Hyperhidrosis: A Prospective Comparative Study. Clinics (Sao Paulo). 2024.
- [Background] 2. Liu X, Wang J, Liu Z, Sun X, Zheng J. Comparison of only T3 and T3-T4 sympathectomy for axillary hyperhidrosis: a retrospective study. J Thorac Dis. 2018;10(4):2095-101.
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Licht PB, Pilegaard HK. Severity of compensatory sweating after thoracoscopic sympathectomy. Ann Thorac Surg. 2004 Aug;78(2):427-31. doi: 10.1016/j.athoracsur.2004.02.087. PMID 15276490